CLINICAL TRIAL: NCT04374734
Title: Automated Quantification of Radiological Pulmonary Involvement in Acute Respiratory Failure
Brief Title: Quantification of Radiological Pulmonary Involvement in Acute Respiratory Failure
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7791
Record Dates: First submitted 2020-04-28; First posted 2020-05-05 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2020-04

CONDITIONS: SARS (Severe Acute Respiratory Syndrome)
Keywords: SARS; Severe Acute Respiratory Syndrome; Automated quantification; Lung volume; Thorax imaging
MeSH Terms: conditions — Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute respiratory failure (ARF) is a common condition and a common reason for urgent medical consultation. Assessing the extent of respiratory impairment is important to improve the management of patients with ARF. When Acute respiratory failure is caused by pathology of the pulmonary parenchyma, quantification of pulmonary radiographic involvement may be a component of the initial assessment of severity. This radiographic quantification would only be usable in clinical routine if it can be automated and provide a real-time result.

The objective of this work is to assess the feasibility of an automated technique for quantifying radiological lung damage in situations of known or potential ARF.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Presenting a situation at risk of acute respiratory failure
* Requiring thorax imaging when they were treated.

Exclusion Criteria:

* Patients with anatomically incomplete thoracic imaging (e.g., technical acquisition error).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presenting a situation at risk of acute respiratory failure
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-04-05 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Retrospective study of the relationship between severe forms of ARF and the extent of lung involvement | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service d' Anesthésie Réanimation Chirurgicale, Strasbourg, France